CLINICAL TRIAL: NCT06452615
Title: Effect of Extracorporeal Shock Wave Therapy on Intercostobrachial Neuralgia Post Mastectomy
Brief Title: Extracorporeal Shock Wave Therapy on Neuropathic Pain Post Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rehab Abutaleb, Faculty of Physical therapy, Department Physical Therapy for Surgery and Burn, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No:P.T.REC/012/004573
Record Dates: First submitted 2024-05-17; First posted 2024-06-11 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Neuropathic Pain
Keywords: Shock Wave Therapy; Mastectomy; Intercostobrachial neuralgia; Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): They will receive Extracorporeal shockwave therapy (ESWT), two session per week for 8 weeks in addition to the routine medical treatment.
  Interventions: Device: Extracorporeal shockwave
- Control group (No Intervention): This group includes thirty female patients suffering from intercostobrachial neuralgia after a modified radical mastectomy. They will receive routine medical treatment.

INTERVENTIONS:
Device: Extracorporeal shockwave — The patients will receive 3000 to 6000 pulses every session by a radius of 15 mm probe (R15) at a frequency of 10 Hz, with energy gradually increasing from 1.4 to 1.5 bar
  Arms: Study group

SUMMARY:
PURPOSE: The main objective of the study is:

to evaluate the therapeutic effect of ESWT on intercostobrachial neuralgia post-mastectomy.

BACKGROUND:

Intercostobrachial neuralgia post-mastectomy is thought to develop from surgical damage to the intercostobrachial nerve, this nerve is injured in 80-100 % of mastectomy patients who undergo axillary lymph nodes dissection.

Pain that is localized in the axilla, medial upper arm, breast, and/or chest wall significantly affects the patient's mood, everyday activities, and social functioning, causing a heavy economic burden on healthcare systems. If poorly treated, patients may develop an immobilized arm, which can lead to severe lymphedema, frozen shoulder syndrome, and complex regional pain syndrome.

HYPOTHESES:

It will be hypothesized that:

Shock wave therapy has no effect in improving intercostobrachial neuralgia post-mastectomy.

DETAILED DESCRIPTION:
Sixty female patients aged 40 and 65 years, suffering from intercostobrachial neuralgia after modified radical mastectomy will be selected from the National Cancer Institute, Cairo, Egypt. They will be randomly assigned into two equal groups, thirty patients each (study group and control group). The intervention in the study group will be conducted for 8 weeks.

Inclusive criteria :

The subject selection will be according to the following criteria:

1. The age range will be from 40 to 65 years.
2. All patients will be female patients suffering from intercostobrachial neuralgia after unilateral modified radical mastectomy.
3. All patients suffering from moderate or severe pain of burning, tingling, numbness, and electric nature persisting for 3-5 months following mastectomy, in the anterior chest wall, axilla, and upper medial arm with altered sensitivity of the skin in the painful area.
4. All patients had unilateral mild to moderate lymphedema (circumference difference 4 cm).
5. All patients will have completed their chemotherapy or radiotherapy treatment.
6. All patients enrolled in the study will have their informed consent.

Exclusive criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Current metastases.
2. Continuing radiotherapy or chemotherapy.
3. History of allergy to coupling agent.
4. Chronic inflammatory diseases and cellulitis.
5. Venous thrombosis.
6. Local infections.
7. Patients with diabetes mellitus (neuritis).
8. Open skin lesions in the painful area.
9. Other causes of arm pain (brachial plexus neuropathy due to radiotherapy, cervical radiculopathy, peri-capsulitis of shoulder joint).

Outcomes:

* ROM of the shoulder joint for flexion and extension
* Level of pain

ELIGIBILITY:
Inclusion Criteria:

1. Age range will be from 40 to 65 years.
2. All patients will be female patients suffering from intercostobrachial neuralgia after unilateral modified radical mastectomy.
3. All patients suffering from moderate or severe pain of burning, tingling, numbness, and electric nature persisting for 3-5 months following mastectomy, in the anterior chest wall, axilla, upper medial arm with altered sensitivity of the skin in the painful area.
4. All patients had unilateral mild to moderate lymphedema (circumference difference 4 cm).
5. All patients will have completed their chemotherapy or radiotherapy treatment.
6. All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

1. Current metastases.
2. Continuing radiotherapy or chemotherapy.
3. History of allergy to coupling agent.
4. Chronic inflammatory diseases and cellulitis.
5. Venous thrombosis.
6. Local infections.
7. Patients with diabetes mellitus (neuritis).
8. Open skin lesions in the painful area.
9. Other causes of arm pain (brachial plexus neuropathy due to radiotherapy, cervical radiculopathy, peri-capsulitis of shoulder joint).

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain | at baseline (pre-treatment), after 4 weeks and after 8 weeks (post-treatment).
  The Visual Analog Scale (VAS) will be used for assessing and quantifying pain exhibited by the patients.
Range of Motion | Measurements will be taken at baseline (pre-treatment), after 4 weeks and after 8 weeks (post-treatment).
  Shoulder Flexion and Abduction will be assessed from supine position

CONTACTS AND LOCATIONS:
Locations (1):
- from the National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No